CLINICAL TRIAL: NCT04177069
Title: Real World Study to Evaluate the Improving Effects of Visucomplex Plus on Quality of Life in Patients With Dry and Wet Age-related Macular Degeneration (AMD)
Brief Title: Evaluate the Improving Effects of Visucomplex Plus on Quality of Life in Patients With AMD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: VISUfarma SpA (Industry)
Responsible Party: Sponsor
Other Study IDs: VF-AMD-VSCLX-2019
Record Dates: First submitted 2019-07-12; First posted 2019-11-26 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: AMD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Visucomplex Plus monotherapy: Patients with early dry AMD will be treated with Visucomplex Plus monotherapy.
  Interventions: Dietary Supplement: Visucomplex Plus
- anti-VEGF drug plus Visucomplex Plus: Dry or wet AMD patients under treatment with a stable dose of an anti-VEGF drug, Visucomplex Plus will be added-on, upon physician decision.
  Interventions: Dietary Supplement: Visucomplex Plus

INTERVENTIONS:
Dietary Supplement: Visucomplex Plus — capsule contains: Lutein, Zeaxanthin, alphalipoic acid MATRIX, Vitamine E, Zinc, Maquibright® (Aristotelian chilensis berry standardized, containing Anthocyanin and delphinidin extracts), Vitamin D and cupper.

SUMMARY:
This is an observational study in which patients affected by dry or wet AMD will be enrolled, after signing the Informed Consent, according to eligibility criteria.

Patients, after signing the Informed Consent, will enter into a screening phase during which the concomitant medication, clinical history, physical examination (including smoking habits) will be checked and the inclusion/exclusion criteria will be assessed.

Then, at the time of Baseline visit (V0) the eligible patients will be given Visucomplex Plus as monotherapy, 1 capsule daily after food, or for dry or wet AMD patients under treatment with a stable dose of an anti-VEGF drug, Visucomplex Plus, 1 capsule daily after food, upon physical decision.

Screening phase and the baseline visit (V0) could coincide.

ELIGIBILITY:
Inclusion Criteria:

* Patient Informed consent form (ICF) signed
* Adult male and female irrespective of their age at the time of the signature of ICF
* Patients affected by dry or wet AMD irrespective of the disease severity and including newly diagnosed patients
* Patients with no treatment for AMD or under treatment with stable doses of anti-VEGF
* Willing to follow all study procedures, including attending all site visits, tests and examinations.

Exclusion Criteria:

* Previously diagnosed optic neuropathies
* Decompensated diabetes or hypertension
* Retinal pathologies including hereditary forms
* Neurological, Neurodegenerative or Cerebrovascular conditions
* Patients with a significantly progressive opacity of lens in the previous 3 months prior to enrolment
* Surgical intervention for cataract in the previous 3 months prior to enrolment
* Previously diagnosed eye inflammatory conditions (uveitis) in the previous 3 months
* Refractive defects beyond the 5 spherical diopters, both positive and negative and over 3 cylindrical
* Any clinically significant history of serious digestive tract, liver, kidney, cardiovascular or hematological disease,
* Known drug and/or alcohol abuse
* Mental incapacity that precludes adequate understanding or cooperation
* Participation in another clinical study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with AMD (dry or wet)
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2019-12-11 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Improvement of QoL in patients affected by AMD (dry or wet) measured through a questionnaire self-administered by the patient partially derived from the VFQ-25, aiming to define a new assessment instrument coupled with the routinely clinical follow up. | measured at baseline and after 4-8 and 12 months of treatment.
  QoL measured through a new questionnaire self-administered

SECONDARY OUTCOMES:
Comparison of improvement scoring of QoL between VFQ-25 and a newly conceived questionnaire | measured at baseline and after 4-8 and 12 months of treatment.
  Comparison of improvement scoring of Quality of Life between the two questionnaires (VFQ-25 and a newly conceived one) at baseline and after 4-8 and 12 months of treatment.
  VFQ-25 is a valid 25-item version of the 51-item National Eye Institute Visual Function Questionnaire (NEI-VFQ).
Visual acuity | measured at baseline and after 4-8 and 12 months of treatment.
  Evaluation of disease progression through Visual acuity.
OCT | measured at baseline and at the end of the observation period (12 months).
  Evaluation of disease progression through Optical Coherence Tomography (OCT).
Questionnaire completion compliance | measured at the end of the observation period (12 months).
  Evaluation of improvement of completion compliance of the new questionnaire versus standard of care one (VFQ-25).
  VFQ-25 is a valid 25-item version of the 51-item National Eye Institute Visual Function Questionnaire (NEI-VFQ).
Likert scales (5 points) | measured at baseline and after 4-8 and 12 months of treatment.
  Evaluation of Patient's treatment judgement and improvement of condition (Likert Scales).
  A Likert scale is a rating scale where patients have to indicate their treatment judgement and improvement of condition crossing a score from 1 to 5.
subject and investigator satisfaction: questionnaire | measured at baseline and after 4-8 and 12 months of treatment.
  Evaluation of subject and investigator satisfaction of the new questionnaire.
  Subject and investigator satisfaction is to be indicated on a scale crossing a score from 1 to 5.

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - Casa di Cura Villa dei Fiori, Acerra, Napoli
  - Ospedale Felice Lotti, Pontedera, Pisa
  - ASST Spedali Civili di Brescia, Brescia
  - Ospedale Policlinico Casilino, Roma

IPD SHARING:
Plan to Share IPD: No